CLINICAL TRIAL: NCT02000193
Title: Maintenance Hormone Therapy With Fulvestrant After First-Line Chemotherapy for Postmenopausal Hormone-receptor-positive (HR) Positive Advanced Breast Cancer: A Multicenter, Prospective Phase II Study
Brief Title: Maintenance Hormone Therapy for Postmenopausal HR Positive Advanced Breast Cancer
Acronym: FANCY
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, wang shusen, professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISSFASL0042
Record Dates: First submitted 2013-11-13; First posted 2013-12-04 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): drug: Fulvestrant treatment : Eligible patients will receive fulvestrant 500 mg intramuscular injection on day 1, 15, 29, then every 28 days.
  The treatment will continue until disease progression or intolerable adverse event
  Interventions: Drug: fulvestrant

INTERVENTIONS:
Drug: fulvestrant — Eligible patients will receive fulvestrant 500 mg intramuscular injection on day 1, 15, and 29， then every 28 days.
  The treatment will continue until disease progression or intolerable AE.
  Other Names: Faslodex

SUMMARY:
This is a prospective, single arm phase II study to evaluate the efficacy and safety of fulvestrant as a maintenance hormone therapy after first-line chemotherapy for postmenopausal HR positive advanced breast cancer.

DETAILED DESCRIPTION:
This is a prospective, single arm phase II study to evaluate the efficacy and safety of fulvestrant as a maintenance hormone therapy after first-line chemotherapy for postmenopausal HR positive advanced breast cancer.

Approximately 58 women who have stable disease or responded to first line chemotherapy with at least 4 and less than 8 weeks of treatment for metastatic breast cancer will be enrolled to this study and receive fulvestrant 500mg as a maintenance therapy. The treatment will continue until the objective disease progression or intolerable AE.

Efficacy will be determined based on tumor assessments performed by each investigator according to RECIST (Response Evaluation Criteria in Solid Tumors ) 1.1. Safety will be monitored based on the frequency and severity of adverse events (AEs), as assessed by Common Terminology Criteria (CTC) grade version 4.0.

Tumor assessments will be assessed by computed tomography (CT) or magnetic resonance imaging (MRI) every 12 weeks for all patients until documented evidence of objective disease progression.

Reporting of SAEs (serious adverse events) to regulatory authorities will be done by the investigator in accordance with local regulations.

ELIGIBILITY:
Inclusion Criteria:

Provision of informed consent Histologically proven HR positive breast cancer

Postmenopausal woman, defined as a woman fulfilling any 1 of the following criteria (based on the NCCN definition of menopause [National Comprehensive Cancer Network 2008]):

Prior bilateral oophorectomy Age ≥60 years Age <60 years and amenorrheic for 12 or more months in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression and follicle stimulating hormone and oestradiol in the postmenopausal range.

Patients have completed first-line chemotherapy for metastatic breast cancer The first-line chemotherapy must be given to patients with visceral disease or progressive disease requiring a fast response Responded(CR or PR) or stabilized(SD>=24 weeks) to first-line chemotherapy for metastatic breast cancer The duration of 1st line chemotherapy for advanced breast cancer had been at least 4 cycles and at most 8 cycles WHO performance status 0, 1 or 2-

Exclusion Criteria:

* Presence of life-threatening metastatic visceral disease, defined as extensive hepatic involvement, or any degree of brain or leptomeningeal involvement (past or present) Prior hormonal treatment for metastatic breast cancer are not allowed More than one line of cytotoxic chemotherapy for metastatic breast cancer Her-2 positive Other malignant tumor (concurrent or previous). Any severe concomitant condition which makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the study protocol, eg, uncontrolled cardiac disease or uncontrolled diabetes mellitus

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-11; Primary Completion 2016-04 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Benefit Rate | 1 year
  defined as the proportion of all treated patients who have a best objective tumour response of CR, PR or SD ≥ 24 weeks

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 1 year
Objective Response Rate(ORR) | 1 year
Number of Participants with Adverse Events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: shusen wang, professor, Principal Investigator — State Key Laboratory of Oncology in South China, Sun Yat-sen University Cancer Center
Locations (1):
- State Key Laboratory of Oncology in South China, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China